CLINICAL TRIAL: NCT06519760
Title: Evaluation of Diagnostic Value of 68Ga-C1 PET/ CT Imaging in Clear Cell Renal Cell Carcinoma
Brief Title: 68Ga-C1 PET/ CT Imaging in Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, GONG Kan, Surgeon, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024#07-17
Record Dates: First submitted 2024-07-17; First posted 2024-07-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Carbonic Anhydrase IX; PET-CT; Clear Cell Renal Cell Carcinoma
Keywords: Carbonic Anhydrase IX; 68Ga-C1; PET-CT; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-C1 (Experimental): Subjects with suspected or confirmed clear cell renal cell carcinoma will receive an intravenous injection of 68Ga-C1 followed by PET imaging. The subjects will also receive a whole-body 18F-FDG PET/CT scan within a one-week period.
  Interventions: Drug: 68Ga-C1

INTERVENTIONS:
Drug: 68Ga-C1 — 68Ga-C1 is injected intravenously with a dose of 0.05-0.10 mCi/kg
  Other Names: CAIX specific PET imaging

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic value of CAIX protein specific probe 68Ga-C1 in PET/CT imaging in clear cell renal cell carcinoma patients. It will also learn about the safety, tolerability and radiation dosimetry of 68Ga-C1.

Researchers will compare the diagnostic value of 68Ga-C1 PET/CT and 18F-FDG PET/CT in Chinese patients with indeterminate renal masses or confirmed clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
Carbonic anhydrase IX (CAIX) is a transmembrane protein which is highly expressed in approximately 95% of clear cell renal cell carcinomas, and it is closely related to tumor progression, patients prognosis and treatment response. Here, we developed a CAIX specific small molecule probe 68Ga-C1, which has shown a good diagnostic accuracy in PET/CT imaging in our preclinical mouse model of clear cell renal cell carcinoma. This enables high-contrast imaging of clear cell renal carcinoma, providing a new imaging method for the precise diagnosis of clear cell renal carcinoma. In this clinical trail, we will compare the diagnostic value of 68Ga-C1 PET/CT and 18F-FDG PET/CT in Chinese patients with indeterminate renal masses or confirmed clear cell renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent；
2. Age ≥18；
3. Patients with confirmed or suspected clear cell renal cell carcinoma;
4. Expected survival ≥6 months.

Exclusion Criteria:

1. Renal mass is known to be a metastasis of another primary tumor;
2. Have other malignancies that require treatment;
3. Have received chemotherapy, radiotherapy, or immunotherapy within 4 weeks;
4. Renal insufficiency with glomerular filtration rate (GFR) ≤ 60 mL/min/1.73 m²;
5. Pregnant and lactating women or female patients plan to become pregnant within 6 months;
6. Uncontrolled psychiatric disorders;
7. Vulnerable population (e.g., being in detention) or have a serious non-malignant disease (e.g., infectious disease, autoimmune disease, or metabolic disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficacy of 68Ga-C1 PET/CT in the evaluation of clear cell renal cell carcinoma | 1 year
  Compare the standardized Uptake Value (SUV) of lesions on 68Ga-C1 and 18F-FDG PET/CT
The diagnostic efficacy of 68Ga-C1 PET/CT in the evaluation of malignant tumors | 1 year
  Compare the number of lesions detected by 68Ga-C1 and 18F-FDG PET/CT, based on the pathology or clinical follow-up as gold standard.

SECONDARY OUTCOMES:
The dosimetry of 68Ga-C1 | 1 year
  Research on the dose distribution of 68Ga-C1 in healthy volunteers and cancer patients by 1-hour dynamic PET/CT acquisition and analyze by the dosimetry software
Quantitative evaluation of 68Ga-C1 | 1 year
  Evaluation of quantitative parameters of 68Ga-C1, such as time-activity curve.
Correlation with pathological expression | 1 year
  Analyze CAIX expression at the imaging level in combination with CAIX expression in pathological specimens

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China